CLINICAL TRIAL: NCT00722293
Title: A Phase I, Open-label, Study of the Safety, Pharmacokinetics, and Pharmacodynamics Dose Escalation of Pazopanib in Combination With Epirubicin or Doxorubicin for Advanced Solid Tumors
Brief Title: A Phase I, Open-label, Study of Pazopanib in Combination With Epirubicin or Doxorubicin for Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEG109603
Record Dates: First submitted 2008-07-23; First posted 2008-07-25 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Neoplasms, Breast
Keywords: Solid tumors; Cancer; Neoplasms, Ovarian; doxorubicin; epirubicin; anti-angiogenesis; pharmacodynamics; pazopanib (GW786034); pharmacokinetics; Soft Tissue; Sarcoma
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Ovarian Neoplasms; Sarcoma | interventions — Doxorubicin; pazopanib; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm A (Experimental): once daily oral administration of pazopanib for Days 1-21 days in combination with epirubicin given as a bolus intravenous administration on Day 3
  Interventions: Drug: Pazopanib (GW786034); Drug: Epirubicin
- Arm B (Experimental): once daily oral administration of pazopanib for Days 1-8 of a 3-week cycle in combination with epirubicin (bolus intravenous administration) on Day 3
  Interventions: Drug: Pazopanib (GW786034); Drug: Epirubicin
- Arm C (Experimental): epirubicin (bolus intravenous administration) on Day 1 with once-daily oral administration of pazopanib for Days 14-21 of a 3-week cycle
  Interventions: Drug: Epirubicin
- Arm D (Experimental): once-daily oral administration of pazopanib (according to schedule selected from either Arm A, B, or C) (3 week cycle) in combination with doxorubicin (bolus intravenous administration) on Day 1 or 3, depending on the schedule selected from either Arm A, B, or C
  Interventions: Drug: Doxorubicin; Drug: Pazopanib (GW786034)

INTERVENTIONS:
Drug: Doxorubicin — Arm D - doxorubicin given as a intravenous bolus injection on Day 1 or Day 3 depending on schedule selected from Arm A, B or C - starting dose 60 mg/m2 and increase to 75mg/m2
  Arms: Arm D
Drug: Pazopanib (GW786034) — Arm A - daily administration of pazopanib on Days 1 through 21 starting at 200mg with a maximum dose of 800mg; Arm B daily administration of pazopanib on Days 1 through 8 of a 3-week cycle starting at 200mg escalating to a maximum dose of 800mg; Arm C daily dose of pazopanib on Days 14 through 21 of a 3-week cycle starting at 200mg escalating to a maximum dose of 800mg; Arm D once daily administration of pazopanib (according to schedule selected from Arm A, B, or C) starting at 400mg escalating to a maximum dose of 800mg
  Arms: Arm A; Arm B; Arm D
Drug: Epirubicin — Arm A and Arm B - epirubicin given as a bolus intravenous injection on Day 3 starting dose 60mg/m2 increase to 90mg/m2 if tolerated; Arm C - epirubicin given as a bolus intravenous injection on Day 1 starting dose 60mg/m2 increase to 90mg/m2 if tolerated
  Other Names: Doxorubicin; Pazopanib (GW786034)
  Arms: Arm A; Arm B; Arm C

SUMMARY:
This is an open-label, four-arm, Phase I, dose escalation study to evaluate the safety and tolerability and to determine the optimal tolerated regimen (OTR) of pazopanib in combination with epirubicin or doxorubicin in patients with advanced solid tumors. Patients will be enrolled in cohorts of 3 to receive escalating doses of pazopanib and epirubicin or doxorubicin. Dose escalation schemas for each study arm are described in the protocol. For each arm, the OTR will be defined as the highest dose combination of the agents where no more than one out of six patients experiences a dose-limiting toxicity. Twelve additional patients in each arm will be studied with the OTR to evaluate toxicity and pharmacokinetics. This will allow an assessment of potential drug-drug interactions. Antitumor activity will be assessed using RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent prior to performance of study specific procedures or assessments, and must be willing to comply with treatment and follow up
* Histologically or cytologically confirmed diagnosis of advanced solid tumor that has failed standard therapy or for which there is no standard therapy and is indicated for treatment with anthracyclines.
* Age greater than or equal to 18 years.
* Adequate organ system function as defined by the protocol.
* ECOG performance value of 0 or 1.
* Less than or equal to one prior line of chemotherapy for advanced disease. Patients with metastatic disease to the brain should have definitive therapy for their brain metastases, should be asymptomatic. (Patients with previously treated brain metastases who are asymptomatic, off steroids and anti-seizure medications for greater than 3 months are eligible for the study).
* There must be measurable disease or evaluable disease for subjects to be included in the cohort expansion phase. Measurable disease is not a criterion for subjects enrolling in the dose escalation phase.
* Has a left ventricular ejection fraction (LVEF) greater than or equal to 50% or greater than or equal to the institution's LLN.
* Women of childbearing potential must have a negative pregnancy test within 2 weeks of starting study drug and use acceptable birth control methods as outlined in the protocol.
* Women may participate if they are of non childbearing potential (bilateral tubal ligation, hysterectomy, post menopausal or bilateral ovariectomy.
* Males with female partners of childbearing potential may participate if they practice acceptable methods of birth control as outlined in the study protocol.
* Able to swallow and retain oral medications.
* Less than or equal to one prior line of chemotherapy for advanced disease.
* Life expectancy of at least 12 weeks.

Exclusion Criteria:

* Prior use of pazopanib or prior treatment with anthracyclines. Prior therapy with other angiogenesis inhibitors is permitted.
* Clinically significant gastrointestinal abnormalities which might interfere with oral dosing.
* Any unstable or serious concurrent condition (e.g., active infection requiring systemic therapy).
* QTc > 480 msecs.
* History of any one or more of the following cardiovascular conditions within the past 6 months:

  * Cardiac angioplasty or stenting
  * Myocardial infarction
  * Unstable angina
  * Symptomatic peripheral vascular disease
  * Class III or IV congestive heart failure
* Any major surgery or trauma within the last 28 days and or presence of non-healing wound, fracture, or ulcer.
* Any unstable or serious concurrent condition.
* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of =140mmHg or diastolic blood pressure (DBP) of = 90mmHg].
* History of cerebrovascular accident (CVA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. Subjects with a recent DVT who have been treated with therapeutic agents (excluding therapeutic warfarin) for at least 6 weeks are eligible.
* Prior major surgery or trauma within 28 days prior to first dose of study drug and /or presence of any non-healing wound, fracture, or ulcer.
* Hemoptysis within 6 weeks prior to first dose of study drug.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with patient's safety, provision of informed consent, or compliance to study procedures.
* Is unable or unwilling to discontinue prohibited medications for 14 days or five half-lives of a drug prior to Visit 1 and for the duration of the study.
* Use of an investigational agent, including an investigational anti-cancer agent, within 28 days or 5 half-lives, whichever is longer, prior to the first dose of study drug.
* Is now undergoing and/or has undergone within 28 days immediately prior to first dose of study drug, any cancer therapy (major surgery, investigational agent, tumor embolization, chemotherapy, radiation therapy, immunotherapy, biological therapy, or hormonal therapy).
* Clinically assessed as having inadequate venous access for PK sampling.
* Lactating and pregnant women should discontinue lactation prior to first use of study drug and refrain from nursing throughout the treatment period and for 14 days after final dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2008-07-08 (Actual); Primary Completion 2012-06-11 (Actual); Study Completion 2014-02-25 (Actual)

PRIMARY OUTCOMES:
Optimum tolerated regimen (OTR) for each combination regimen in each arm of the study.OTR determined by evaluation of AEs and change in lab values.OTR defined as highest dosing regimen that results in dose limiting toxicity in no more than 1 of 6 subject | Subjects will continue on the study until disease progression occurs or one of the discontinuation criteria is met up to approximately 48 months.

SECONDARY OUTCOMES:
Safety assessments, including routine physical exam findings, vital signs, clinical laboratory tests (chemistry and hematology to include coagulation factors), clinical monitoring and/or observation, and adverse event reporting. | Safety assessment timing is noted on the Time and Events Table. Subjects will continue on the study until disease progression occurs or one of the discontinuation criteria is met up to approximately 48 months.
Safety and tolerability endpoints will include cardiac function (left ventricular ejection fraction) monitored by either MUGA or ECHO. A 12-lead ECG will also be monitored. | Safety assessment timing is noted on the Time and Events Table. Subjects will continue on the study until disease progression occurs or one of the discontinuation criteria is met up to approximately 48 months.
Pharmacokinetic endpoints will be AUC, Cmax, Tmax, and t1/2 of pazopanib, epirubicin, and doxorubicin, and clearance of epirubicin and doxorubicin if data are sufficient. | PK samples will only be collected in Cycle 1 and Cycle 2. Subjects will continue on the study until disease progression occurs or one of the discontinuation criteria is met up to approximately 48 months.
Assessment of anti-tumor activity using RECIST criteria will be recorded as complete response, partial response, stable disease, or progressive disease. | Subjects will continue on the study until disease progression occurs or one of the discontinuation criteria is met up to approximately 48 months.
Levels of circulating cytokine and angiogenic factors (CAF) biomarkers (such as IL 2, IL-10, VEGF, sVEGFR2) in plasma will be determined. | Biomarker samples will only be collected in Cycles 1, 2, and 3. Subjects will continue on the study until disease progression occurs or one of the discontinuation criteria is met up to approximately 48 months.
Assessment of circulating BMD angiogenic cells in cancer peripheral blood in patients before and during treatment with oral pazopanib (continuous and intermittent regimens) and epirubicin or doxorubicin. | Biomarker samples will only be collected in Cycles 1 and 2. Subjects will continue on the study until disease progression occurs or one of the discontinuation criteria is met up to approximately 48 months.
Gene expression profiling in selected subpopulations of BMD angiogenic cells in peripheral blood of cancer patients before and during treatment with pazopanib (continuous or intermittent regimens) in combination with epirubicin or doxorubicin. | Biomarker samples will only be collected in Cycles 1 and 2. Subjects will continue on the study until disease progression occurs or one of the discontinuation criteria is met up to approximately 48 months.
Genetic variants in candidate genes in the host DNA will be evaluated | One pharmacogenetic sample will be collected during the study ideally in Cycle 1. Subjects will continue on the study until disease progression occurs or one of the discontinuation criteria is met up to approximately 48 months.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- GSK Investigational Site, Milan, Lombardy, Italy
- Switzerland (3):
  - GSK Investigational Site, Bellinzona
  - GSK Investigational Site, Lausanne
  - GSK Investigational Site, Sankt Gallen

REFERENCES:
- See also: Results for study VEG109603 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/VEG109603?search=study&search_terms=VEG109603#rs